CLINICAL TRIAL: NCT05395507
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial of Pegylated Interferon Alfa-2b Versus Interferon Alfa Therapy in the Treatment of Adult Essential Thrombocythemia
Brief Title: Pegylated Interferon Alfa-2b Versus Interferon Alfa Therapy in Adult Essential Thrombocythemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022004
Record Dates: First submitted 2022-05-10; First posted 2022-05-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-11

CONDITIONS: Essential Thrombocytopenia
Keywords: Essential Thrombocytopenia; Interferon Alfa; Pegylated Interferon Alfa-2b; Efficacy; Safety
MeSH Terms: interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Interferon Alpha (Active Comparator): Recombinant Interferon Alpha, with an initial dose of 300 wu three times a week. Other interferons that have been listed can be used if Recombinant Interferon Alpha (300 wu) is not available.
  Interventions: Drug: Recombinant Interferon Alpha
- Pegylated Interferon Alfa-2b (Experimental): Pegylated Interferon Alfa-2b, with an initial dose of 135 ug at week 0 , and then 180 ug once a week from week 1 to week 52.
  Interventions: Drug: Pegylated interferon alfa-2b

INTERVENTIONS:
Drug: Recombinant Interferon Alpha — Recombinant Interferon Alpha, with an initial dose of 300 wu three times a week. Other interferons that have been listed can be used if Recombinant Interferon Alpha (300 wu) is not available.
  Arms: Recombinant Interferon Alpha
Drug: Pegylated interferon alfa-2b — Pegylated Interferon Alfa-2b, with an initial dose of 135 ug at week 0 , and then 180 ug once a week from week 1 to week 52.
  Arms: Pegylated Interferon Alfa-2b

SUMMARY:
Objectives: To compare the efficacy and safety in Adult patients (≥18 years) diagnosed as essential thrombocythemia treated with the Pegylated Interferon Alfa-2b vs. Interferon Alfa. Study Design: A prospective, open-label, multicenter, randomized controlled clinical trial.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, randomized controlled clinical trial between Interferon Alfa and Pegylated Interferon Alfa-2b in adult essential thrombocythemia (≥18 years).

Patients will be randomly divided into the following two treatment groups: 1. Recombinant Interferon Alpha, with an initial dose of 300 wu three times a week. Other interferons that have been listed can be used if Recombinant Interferon Alpha (300 wu) is not available. 2. Pegylated Interferon Alfa-2b, with an initial dose of 135 ug at week 0 , and then 180 ug once a week from week 1 to week 52.

The dosage will be adjusted according to the results of laboratory examinations and patient tolerance. The patient will be transferred to the other group if intolerance or resistance occurs.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Male or Female.
* Diagnosis of essential thrombocythemia according to the 2016 World Health Organization criteria.
* Those who have not use interferon within 4 weeks before the first medication.
* Patients with indications for cytoreductive therapy.
* Men and women with reproductive potential, as well as all women with menopause less than 2 years, must agree to use acceptable contraceptive methods until 28 days after the last dose of study drug, and women must agree not to breastfeed during the study period.
* Voluntary written informed consent.

Exclusion Criteria:

* Resistance, or intolerance, or any contraindications to interferon.
* Patients with active thrombosis or active bleeding.
* Neutrophil count < 1.0x10^9/L.
* Hemoglobin < 11g/dL for male, or < 10g/dL for female.
* Poor control of thyroid dysfunction.
* Patients with a prior malignancy within the last 3 years.
* Patients with severe cardiac or pulmonary dysfunction.
* Severe renal damage (creatinine clearance < 30 ml / min).
* Severe liver dysfunction (ALT or AST > 2.5×ULN).
* Patients with hepatitis B virus, hepatitis C virus replication or HIV infection.
* Patients with a history of drug / alcohol abuse (within 2 years before the study).
* Patients that have participated in other experimental researches within one month before enrollment.
* History of psychiatric disorder.
* Any other circumstances that the investigator considers that the patient is not suitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete hematological remission (CHR) rates | From the start of study treatment (Week 0) up to the end of Week 52
  The CHR rates defined as European Leukemia Net will be compared between the two groups.

SECONDARY OUTCOMES:
CHR rates at week 24 and 36 | From the start of study treatment (Week 0) up to the end of Week 24 and Week 36, respectively
  The CHR rates at week 24 and 36 will be compared between the two groups
Time to CHR | From the start of study treatment (Week 0) up to the end of Week 52.
  The time of reaching CHR will be compared between the two groups
The proportion of patients crossed to the contralateral group | From the start of study treatment (Week 0) up to the end of Week 52.
  The proportion of patients crossed to the contralateral group will be compared between the two groups
The CHR rates after crossover | From the start of study treatment (Week 0) up to the end of Week 52.
  The CHR rates within 52 weeks after crossover
Impact of therapy on driver mutations | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the proportion of subjects that display change on key biomarkers of the disease- JAK2V617F, CALR, MPL mutations.
Impact of therapy on non-driver mutations | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the proportion of subjects that display change on key non-driver biomarkers of the disease-DNMT3A, ASXL1, TET2 or other mutations.
Change of splenomegaly | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the proportion of subject with improvement and no progress rate of splenomegaly between the two groups.
Change of bone marrow pathology | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the rate of patients with improvement and no progress rate of bone marrow pathology between the two groups
The incidence of major thrombotic events | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the incidence of major thrombotic events between the two groups.
The incidence of major bleeding events | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the incidence of major bleeding events between the two groups.
The incidence of progressing to bone marrow fibrosis | From the start of study treatment (Week 0) up to the end of Week 52.
  The incidence of progressing to bone marrow fibrosis will be compared between the two groups
The incidence of progressing to acute leukemia | From the start of study treatment (Week 0) up to the end of Week 52.
  The incidence of progressing to acute leukemia will be compared between the two groups
Change in Myeloproliferative Neoplasm Symptom Assessment Form total symptom score | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the proportion of subjects that display change in Myeloproliferative Neoplasm Symptom Assessment Form total symptom score (0-100 scores, higher scores mean a worse outcome) between different treatment groups.
Change of quality of life | From the start of study treatment (Week 0) up to the end of Week 52.
  Compare the rate of patients with improvement in quality of life between the two groups (assessed by EORTC quality of life scale QLQ-C30 V3.0 questionnaire).
Change of microcirculation disturbance | From the start of study treatment (Week 0) up to the end of Week 52.
  The rate of patients with improvement in microcirculation disturbance (such as pruritus, headache, dizziness, chest tightness, erythematous limb pain and limb paresthesia) will be compared between the two groups
Specific pre-defined toxicity | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare incidence of specific pre-defined toxicity including fatigue, flu-like symptoms, dizziness, injection site necrosis, dyspnea, pain, depression, blurred Vision, insomnia, anorexia, weight Loss, weakness, pruritis, sweating, fever, decreased Libido, hot Flashes, flushing.

OTHER OUTCOMES:
Changes of immune cell subgroups | From the start of study treatment (Week 0) up to the end of Week 52.
  The proportion of T lymphocyte, B lymphocyte and dendritic cell subsets and the changes of gene expression profile of these cells will be analyzed before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Rongfeng Fu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Rong Fu, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China